CLINICAL TRIAL: NCT06697223
Title: A Randomized, Multi-center, Controlled, In Vivo Study to Assess the Recovery and Survival of Radiolabeled Autologous Apheresis Platelet Components Suspended in 100% Plasma Treated With the INTERCEPT Blood System for Platelets With LED Illuminator Stored for 5 Days
Brief Title: A Study to Assess Recovery and Survival of Radiolabeled Apheresis Platelet Components Treated With the INTERCEPT Blood System for Platelets With LED Illuminator.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLI 00183
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-01

CONDITIONS: Healthy Subjects
Keywords: INTERCEPT; Recovery; 5 Days; Survival; Radiolabel; Autologous; LED Illuminator; Apheresis Platelets
MeSH Terms: interventions — Platelet Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Simultaneous administration of Test and Control platelets (Other): INTERCEPT treated platelets (Test) from 24 healthy subjects, stored for 5 days, will be prepared for radiolabeling following the Variant 1 methodology. The radiolabeled autologous Test and Control platelets, approximately 5 to 30 mL, will be simultaneously administered intravenously into the subject.
  Interventions: Device: INTERCEPT Blood System for Platelets with LED Illuminator

INTERVENTIONS:
Device: INTERCEPT Blood System for Platelets with LED Illuminator — Apheresis platelet components in 100% plasma collected using the Trima separator, prepared with the INTERCEPT Blood System for Platelets (Test Platelets) using the LED Illuminator and stored for 5 days at 20 to 24°C with continuous agitation.

SUMMARY:
The objective of this study is to assess the post-infusion recovery and survival of platelets in 100% Plasma treated with INTERCEPT Blood System for Platelets with LED Illuminator and stored for 5 days after apheresis collection. The post-infusion recovery and survival of autologous radiolabeled 5-day INTERCEPT platelets (Test) stored in 100% plasma will be measured in comparison to fresh autologous radiolabeled platelets (Control).

DETAILED DESCRIPTION:
The study population will consist of healthy subjects who meet the FDA, AABB, and site-specific research donor eligibility criteria for an apheresis platelet collection.

Apheresis platelets (single or double) will be collected in 100% plasma on the Trima Accel® Automated Blood Collection system. Each study apheresis collection will be processed using the INTERCEPT Blood System for Platelets; apheresis platelets containing a platelet dose of 4.0 to 5.2 x10^11 platelets in 300 to 390 mL of plasma will be processed using the INTERCEPT Large Volume (LV) processing set. The INTERCEPT process will begin on either the day of collection (Day 0) or the day following collection (Day 1); illumination must occur within 24 hours after the end of collection. Test platelet components will be stored for up to 5 days, after collection, in 100% plasma.

At the end of storage, an aliquot of Test platelets will be aseptically removed from each subject's INTERCEPT platelet storage container and prepared for radiolabeling. Samples for in vitro platelet testing will be collected prior to INTERCEPT treatment (Day 0/1), post INTERCEPT treatment (Day 1/2), and at the end of storage (Day 5).

The recovery and survival for Test platelets will be compared against the fresh platelet Control. Recovery and survival of INTERCEPT platelets will be assessed after 5 days of storage for up to 24 evaluable subjects.

Test and Control platelets will be randomly radiolabeled with either 51Cr as sodium radiochromate (Na251CrO4) or 111In as Indium Oxine, depending upon randomization. Subjects will be randomized with equal probability to the radiolabeling sequences (111In/51Cr vs. 51Cr/111In) for Test INTERCEPT platelets/Control fresh platelets. After radiolabeling, the autologous Control and Test platelet samples will be simultaneously infused into the subject.

Blood samples will be drawn immediately before infusion and for radioactivity measurements at 2 hours ±15 min post-infusion (Day 0), and 6 more samples will be drawn at 1 (within ±4 hours from time of infusion), 2, 3, 5±1, 7/8, and 11±1 days post-infusion (DPI)). The exact time of each sample draw will be recorded.

Subjects will be monitored for safety (adverse events including transfusion reactions) from the time of the apheresis procedure until 24 hours after the last DPI blood sample is drawn.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Normal health status (as determined by the Investigator review of medical history and blood donor physical exam)
* Complete blood count (CBC) and serum chemistry values within normal limits or outside of normal reference range but determined by the Investigator, and consultation with the Sponsor, to be not clinically significant.
* Meet FDA, AABB or institutional guidelines for allogeneic and plateletpheresis donor qualifications with the following exceptions:

  o Deferrals due to travel, tattoos/piercings, male to male sexual contact as institutional policies allow
* All routine infectious disease testing must be negative or non-reactive (during screening)
* Subjects of childbearing potential must agree to use a medically acceptable (as per the Investigator) method of contraception throughout the study
* Signed and dated informed consent form

Exclusion Criteria:

* Clinically significant acute or chronic disease (as determined by the Investigator)
* Treatment with aspirin or aspirin-containing medications within 7 days of apheresis or treatment with non-steroidal anti-inflammatory drugs (NSAID), anti-platelet agents or other drugs affecting platelet viability within 3 days of apheresis (e.g., ibuprofen or other NSAIDs)
* Subject received platelet inhibitors within 14 days of donation (e.g., clopidogrel, ticlopidine, amphetamines (e.g., Adderall, Dexedrine))
* Immunosuppressive therapy (e.g., oral or IV prednisone) within the past 28 days
* Treatment with any medication known to affect platelet viability
* Pregnant or nursing females
* Received an investigational drug within the past 28 days or current participation in another clinical interventional study
* Non study blood component donation throughout the study
* Subjects with positive cocaine and/or amphetamine result from urine drug screen.
* Splenectomized subjects
* History of known hypersensitivity to 51Chromium or 111Indium

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Post infusion recovery of Test platelets at end of 5 day storage | After 5 Day Storage
Post infusion survival of Test platelets at end of 5 Day storage | After 5 Day Storage

SECONDARY OUTCOMES:
Platelet Dose in Test Component: Percentage of Test components with ≥ 3.0×10^11 platelets | At the end of INTERCEPT treatment on Day 1 or Day 2
Platelet Yield Retention in Test Component: Percentage of Test components with ≥80% platelet yield retention | At the end of INTERCEPT treatment on Day 1 or Day 2
pH 22°C of Test Component: Percentage of Test components with pH 22°C ≥ 6.2 | At end of 5 Day storage

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - American Red Cross Research Laboratory, Norfolk, Virginia
  - Bloodworks Northwest Research Institute, Seattle, Washington